CLINICAL TRIAL: NCT07231536
Title: Investigating Dual-Model Effects of Acute Pre-Class Physical Exercise on Inhibitory Control: A Cluster-Randomized Classroom Trial
Brief Title: Boosting Executive Function With Real-class Exercise
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shenzhen University (Other)
Responsible Party: Principal Investigator, Liye Zou, Professor, Shenzhen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: ShenzhenURealClassExercise
Record Dates: First submitted 2025-11-13; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Executive Functions (EF)
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- mentally passive sedentary behavior (No Intervention)
- mentally active sedentary behavior (Active Comparator)
  Interventions: Behavioral: Mentally active sitting
- 5-minute physical exercise (Experimental)
  Interventions: Behavioral: 5-minute physical exercise
- 10-minute physical exercise (Experimental)
  Interventions: Behavioral: 10-minute physical exercise

INTERVENTIONS:
Behavioral: Mentally active sitting — Participants remain seated for approximately 10 minutes before class while engaging in a cognitively stimulating activity designed to elicit mental effort without physical exertion.
  Arms: mentally active sedentary behavior
Behavioral: 5-minute physical exercise — Participants remain seated quietly for approximately 5 minutes before class without performing any structured cognitive or physical tasks. Then they will have 5-minute physical exercise before class.
  Arms: 5-minute physical exercise
Behavioral: 10-minute physical exercise — Participants do 10-minute physical exercise before class.
  Arms: 10-minute physical exercise

SUMMARY:
The goal of this study is to examine the effects of acute pre-class physical exercise on executive function in real classroom settings. The main question it aims to answer is, "Does acute pre-class exercise enhance executive function compared to sedentary conditions?" Participants were students from primary school assigned by class to engage in one of several pre-class conditions: mentally passive sitting, mentally active sitting, 5-minute physical exercise, or 10-minute physical exercise. A cluster-randomized trial design was used to ensure ecological validity in authentic classroom environments. Cognitive tasks measuring inhibitory control were administered at baseline and pre-/post-class.

The results indicate that pre-class exercise leads to greater improvements in inhibitory control than sedentary conditions, suggesting that integrating brief exercise sessions before lessons may be an effective strategy to optimize learning in educational contexts.

ELIGIBILITY:
Inclusion Criteria:

* right-handed, had normal or corrected-to-normal visual acuity, and normal color vision

Exclusion Criteria:

* reported a history of cardiovascular, metabolic, gastrointestinal, neurological, or psychiatric disorders or conditions requiring medical attention.

Ages: 9 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 240 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-05-17 (Estimated); Study Completion 2026-06-16 (Estimated)

PRIMARY OUTCOMES:
Domain- specific Cognition | Measurements were taken at three time points: baseline (0:00), after the 10-minute intervention (0:15), and following the 40-minute class (0:60).
  This indicator is measured using the computerized Children's Version of the math-related Negative Priming task. The underlying measures employed are task accuracy and reaction time, without involving any physiological measurements.
Domain-general Cognition | Measurements were taken at three time points: baseline (0:00), after the 10-minute intervention (0:15), and following the 40-minute class (0:60).
  This indicator is measured using the computerized Children's Version of the Erikson Flanker task. The underlying measures employed are task accuracy and reaction time, without involving any physiological measurements.